CLINICAL TRIAL: NCT07266532
Title: Evaluation of the Safety and Efficacy of Topical Application of Lactobacillus Crispatuson the Forearm for Treating Obesity-Induced Skin Barrier Dysfunction: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Topical Lactobacillus Crispatus for Skin Barrier Dysfunction in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LL-KY-2025229-02
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Skin Barrier to Water Loss; Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical L. crispatus Treatment Group (Experimental)
  Interventions: Biological: Topical L. crispatus Treatment Group
- Topical Inactivated Lactobacillus crispatus Application Group (Sham Comparator)
  Interventions: Biological: Topical Inactivated Lactobacillus crispatus Application Group

INTERVENTIONS:
Biological: Topical Inactivated Lactobacillus crispatus Application Group — Once daily, 3mL of inactive Lactobacillus crispatus solution was applied to the bilateral forearms at a diameter of 3cm 10cm from the carpal wrinkles
  Arms: Topical Inactivated Lactobacillus crispatus Application Group
Biological: Topical L. crispatus Treatment Group — Once daily, 3mL of Lactobacillus crispatus solution was applied to the bilateral forearms at a diameter of 3cm 10cm from the carpal wrinkles
  Arms: Topical L. crispatus Treatment Group

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of topical application of Lactobacillus crispatuson the forearm for treating obesity-induced skin barrier impairment in individuals aged 18-45 with BMI ≥25. The study focuses on the following questions:

Can topical application of Lactobacillus crispatusreduce skin barrier damage, as measured by transepidermal water loss (TEWL), in obese participants?

Does modulation of the skin microbiota with Lactobacillus crispatusimprove skin barrier function, hydration, and reduce local inflammation?

Is the topical intervention safe and well-tolerated, with minimal adverse effects?

Preliminary data from obese volunteers and mouse models revealed significantly elevated TEWL and reduced Lactobacillusabundance in the skin microbiome of obese individuals, supporting the investigation of probiotic restoration.

Researchers will compare outcomes across two groups:

Intervention Group (Obese) : Daily topical application of active Lactobacillus crispatussolution (1×10⁷ CFU in 3 mL) to a 3-cm diameter area on both forearms.

Placebo Control Group (Obese) : Daily topical application of inactivated Lactobacillus crispatussolution (identical appearance and volume).

Participant Procedures:

Apply the assigned topical solution daily to the forearm for 4 weeks.

Undergo non-invasive skin testing, including TEWL measurements and skin hydration assessments, at baseline and study completion (Week 4).

Provide skin swab samples at baseline and Week 4 for microbiome analysis (16S rRNA sequencing) and inflammation marker detection (e.g., IL-1β, TNF-α via ELISA).

Complete weekly check-ins to report adverse effects (e.g., skin irritation, erythema) and adherence, with follow-ups at Weeks 1, 2, and 3.

Maintain a daily electronic or paper diary to record application time, dose, and any skin reactions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Meets 2020 WHO BMI classification:
* a. Normal weight (18.5-24.9 kg/m²)
* b. Overweight (25-29.9 kg/m²)
* c. Obesity (≥30 kg/m²)
* 2. Presence of skin barrier impairment (e.g., dryness, erythema, desquamation, or itching)
* 3. Age 18-40 years
* 4. Generally good health (no active systemic diseases)
* 5. Able and willing to provide written informed consent
* 6. No use of oral/topical medications or probiotics within 6 months prior
* 7. No active skin disease or traumatic skin lesions

Exclusion Criteria:

* 1. Known allergy or hypersensitivity to probiotics, placebo, or investigational product
* 2. Active skin disease (e.g., psoriasis, eczema, infection) requiring treatment
* 3. Severe medical conditions:
* a. Cardiopulmonary disease (NYHA class III/IV)
* b. Uncontrolled diabetes (HbA1c >9%)
* c. Autoimmune disorders
* 4. Pregnant or breastfeeding women
* 5. Any condition that may interfere with protocol compliance (per investigator judgement), including:
* a. Inability to understand study procedures
* b. History of poor clinical trial adherence
* 6. Concurrent participation in other interventional trials

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2025-12-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Mean change in transepidermal water loss (TEWL, g/h/m²) on the volar forearm from baseline to 1 month after intervention, measured by Tewameter | Baseline through 1 month after intervention
  TEWL will be assessed on the volar aspect of the forearm using a Tewameter device under standardized environmental conditions (controlled temperature and humidity). At each time point, TEWL will be measured at three predefined skin sites on the volar forearm, and the average value will be used. The primary outcome will be the mean change in TEWL (g/h/m²) from baseline (Day 0) to 1 month after intervention. Lower TEWL values indicate improved skin barrier function.

SECONDARY OUTCOMES:
Change in skin hydration measured by Corneometer | Baseline through 1 month after intervention
  Skin hydration will be assessed using a Corneometer device. Outcomes will be expressed as mean skin capacitance values (arbitrary units) at baseline and post-intervention.
Change in clinical skin health score | Baseline through 1 month after intervention
  Skin dryness, scaling, erythema, itching, and allergy-related symptoms will be evaluated using a standardized Skin Dryness Scoring System. Data will be reported as mean score change from baseline.
Change in body weight and BMI | Baseline through 1 month after intervention
  Participants' body weight (kg) and BMI (kg/m²) will be recorded at baseline and post-intervention. Data will be reported as mean change.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No